CLINICAL TRIAL: NCT03437148
Title: Shunt Quantification in Atrial Septal Defect Using Inert Gas Rebreathing and Thoracic Bioimpedance: Comparison With the Gold Standard Method
Brief Title: Non-Invasive Shunt Quantification in Interatrial Communication
Acronym: NISQIC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulty
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Sport Medicine Department, CHU Clermont-Ferrand (Unknown); Cardiology and Vascular Department, CHU Clermont-Ferrand (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHU-373; 2017-A03149-44 (Other: 2017-A03149-44)
Record Dates: First submitted 2018-01-31; First posted 2018-02-19 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Congenital Heart Diseases; Hemodynamic; Cardiac Output
Keywords: Pulmonary to systemic blood flow; Non-invasive measurement; Inert gas rebreathing; Bioimpedance cardiograph; Atrial Septal Defect; Congenital heart disease; Cardiac Output
MeSH Terms: conditions — Heart Defects, Congenital; Heart Septal Defects, Atrial

STUDY DESIGN:
Masking Description: NO MASKING
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with Atrial septal defect type Ostium Secundum (Experimental): patients with Atrial septal defect type Ostium Secundum, eligible for an interventional closure
  Interventions: Device: Innocor®; Device: Physioflow®

INTERVENTIONS:
Device: Innocor® — Inert gas rebreathing device: Innocor® (Innovision, Odense, Denmark)
Device: Physioflow® — Bioimpedance cardiograph: Physioflow® (Manatec, France)

SUMMARY:
Shunt quantification in atrial septal defect (ASD) is estimated by Echocardiography-Doppler, with the pulmonary-to-systemic blood flow ratio: Qp/Qs. Higher is the ratio, more important is the shunt, and the consequence on right ventricular function. A value higher than 1.5 is one of the criteria for percutaneous closure of Secundum ASD. Maatouk and al. have demonstrated that a shunt fraction (Qp/Qs) over 3 is a predictive factor of an incomplete reversibility of the right ventricular remodeling [1]. Even if the accuracy of Doppler echocardiography is admitted for Qp/Qs measurement, there is still some technical difficulties. Thus, the right cardiac catheterization for O2 consumption measurement by the direct Fick method is used. The major inconvenient is the potential risk of adverse effects. Non-invasive methods have been developed using physical properties (as the thoracic bioimpedance) or inert gas rebreathing technique. Thoracic Bioimpedance (TB) and inert gas rebreathing (IGR) techniques have been studies on healthy individual and different respiratory or cardiac diseases to evaluate the cardiac output (CO). TB and IGR measure the systemic and pulmonary blood flow respectively. Without shunt the pulmonary blood flow is equal to the systemic blood flow.

Thus, Investigator suppose that combine the two techniques in disease with shunt, will allow a quantification of the shunt fraction Qp/Qs as accurate as with the gold standard technique (Fick method and Echocardiography Doppler).

The purpose of the study is to evaluate the feasibility and the accuracy of the non-invasive measurement of the Qp/Qs ratio in secundum ASD using the IGR technique and the TB versus the two gold standard techniques: the Fick method and the Echocardiography-Doppler.

The study hypothesizes that the values of Qp et Qs determined by IGR et TB respectively are in the same range of values that the one determined by gold standard techniques.

DETAILED DESCRIPTION:
Shunt quantification and their hemodynamic consequences have a major importance in the evaluation of heart diseases. Atrial septal defect (ASD) has an intracardiac left-to right shunt, leading to an over pulmonary output with ventricular and pulmonary effects. Measurements of the LTR in ASD requires the determination of the pulmonary blood flow (Qp) and the systemic blood flow (Qs).

Two gold standard techniques are usually used to measure the pulmonary to systemic blood flow ratio (Qp/Qs): either invasive by performing a right heart catheterization, with the direct Fick method, or non-invasive by using the Echocardiography-Doppler (ED) First determine by ED by the successively measure of the Qp at the pulmonary annular and the Qs at the aortic annular, this technique is largely available, reproducible and accurate.

However, some limits are pointed with this non-invasive gold standard method: underestimation of shunt quantification in case of large septal defect, the accuracy depends on the operator experience, the lack of precision to measure pulmonary annular area especially on adults leading to a wrong measure of the pulmonary blood flow.

In case of doubt about pulmonary hypertension or difficulties in hemodynamic evaluation, the cardiologists perform a right heart catheterization to measure the CO by the Fick method .

Concerning the other non-invasive approach, thoracic bioimpedance (TB) have been developed in the middle of the twenty-one centuries by Kubiceck to measure cardiovascular parameters in astronauts has been largely study. Moreover, hemodynamic parameters are not stable but varies continuously according to the "hemodynamic state".

High of interest in the field of the non-invasive hemodynamic device, Inert gas rebreathing (IGR) measures the pulmonary blood flow, at rest and on exercise in healthy patient and different cardiorespiratory diseases. The Innocor® (Innovision, Odense, Denmark) uses a rebreathing bag containing a mixing of N2O (0,5%) SF6 (0,1%) and O2 (28%) diluted with atmospheric air. At the steady state of the insoluble inert gas, sulphur hexafluoride SF6, the wash out rate of N2O during rebreathing is calculated, which is proportional to the Qp. Many studies on healthy people confirms its accuracy, safety, reproducibility to measure CO . Agostoni et al. assess the Innocor® on patients with stable heart failure at rest and exercise comparatively to Thermodilution (ThD) and Fick method . They found a good correlation between the three methods at exercise. They found a tendency on underestimation of the IGR technique for CO measurement in comparison to Fick method . Few studies are available on the IGR technique use in CHD population. Tested on a paediatric population, investigators have proved its feasibility on exercise.Secondary they focused on ASD paediatric population. The CO were measured at exercise before and after percutaneous or surgical closured. They confirm the reproducibility, and feasibility of the IGR . Investigators found a similar agreement with the Fick method for patients with CHD without shunting or with right-to-left shunt .

To our knowledge, no study has focused on the concomitant used of two non-invasive technique to measure the shunt fraction in diseases with shunt. Some have suggested the interest of such a method in chronic obstructive pulmonary disease (COPD) .In fact, CO measured at rest and exercise shows a statistical difference between the IGR and TB due to the shunt effect and right-to-left shunt in COPD. Thus, the IGR and TB determine a pulmonary cardiac output (Qp) and a systemic cardiac output (Qs) respectively.

Based on these results, Investigator hypothesis that the combined used of the IGR and TB will enhance the precision and accuracy of the shunt fraction measurement.

The aim of this study is to validate the double non-invasive pulmonary-to-systemic ratio measurements on ostium secundum ASD in comparison to the two-gold standard method: the direct Fick method and the Echocardiography-Doppler.

ELIGIBILITY:
Inclusion Criteria:

* cooperate patients over 18 years, having a OS ASD with an indication of interventional closure according to the European Cardiology society guidelines of 2010.
* Patients with significant shunt (signs of right ventricular volume overload) and Pulmonary Vascular Resistance (PVR) <5WU
* ASD, regardless the size, with suspicion of paradoxal embolism
* Patients with PVR > or egal 5 WU but <2/3 Systemic Vascular Resistance or Pulmonary Arterial Pressure < 2/3 systemic pressure and evidence of net Left-to Right shunt (Qp/Qs > 1,5)
* with the French Social Security System

Exclusion Criteria:

* Pregnant women and breastfeeding women
* Difficulties of cooperation (patient under assisted ventilation)
* Chronic Obstructive Pulmonary disease or respiratory failure
* Complex congenital heart disease
* Antiplatelet contraindication
* Patients under protection, vulnerable patients
* No consent
* Contraindication of the non-invasive devices
* Physioflow (Manatec, France): patients with pacemaker, with a cardiorespiratory support and assistance, severe aortic insufficiency
* Innocor (Innovision, Odense, Denmark): to our knowledge, and according to the user instructions, there is no contraindication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-10-03 (Actual)

PRIMARY OUTCOMES:
shunt fraction | at 1 hour
  Accuracy of Qp/Qs ratio measurements by the double non-invasive technique and the gold standard method (non-invasive: Echocardiography Doppler; invasive: direct Fick method) before interventional closure of ASD

SECONDARY OUTCOMES:
shunt fraction Qp/Qs after closure | at 1 hour
  Qp/Qs measurements by the double non-invasive technique in comparison to Echocardiography-Doppler after interventional closure

CONTACTS AND LOCATIONS:
Overall Officials: Ruddy RICHARD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Background] Maatouk F, Ben Farhat M, Betbout F, Gamra H, Ben Hamda K, Jarrar M, Hammami S, Added F, Ben Gadha N, Dridi Z. [Right ventricular dilatation and intraventricular septal motion after surgical closure of atrial septal defect]. Arch Mal Coeur Vaiss. 2001 Mar;94(3):204-10. French. PMID 11338255
- [Background] Okamoto M, Miyatake K, Kinoshita N, Nakasone I, Ohwa M, Takao S, Fusejima K, Sakakibara H, Nimura Y. [Noninvasive determination of the ratio of pulmonary to systemic blood flow with two-dimensional Doppler echocardiography: efficacy and limitation]. J Cardiogr. 1984 Jun;14(1):189-200. Japanese. PMID 6520422
- [Background] Sanders SP, Yeager S, Williams RG. Measurement of systemic and pulmonary blood flow and QP/QS ratio using Doppler and two-dimensional echocardiography. Am J Cardiol. 1983 Mar 15;51(6):952-6. doi: 10.1016/s0002-9149(83)80172-6. PMID 6829471
- [Background] Baumgartner H, Bonhoeffer P, De Groot NM, de Haan F, Deanfield JE, Galie N, Gatzoulis MA, Gohlke-Baerwolf C, Kaemmerer H, Kilner P, Meijboom F, Mulder BJ, Oechslin E, Oliver JM, Serraf A, Szatmari A, Thaulow E, Vouhe PR, Walma E; Task Force on the Management of Grown-up Congenital Heart Disease of the European Society of Cardiology (ESC); Association for European Paediatric Cardiology (AEPC); ESC Committee for Practice Guidelines (CPG). ESC Guidelines for the management of grown-up congenital heart disease (new version 2010). Eur Heart J. 2010 Dec;31(23):2915-57. doi: 10.1093/eurheartj/ehq249. Epub 2010 Aug 27. No abstract available. PMID 20801927
- [Background] Kubicek WG, Karnegis JN, Patterson RP, Witsoe DA, Mattson RH. Development and evaluation of an impedance cardiac output system. Aerosp Med. 1966 Dec;37(12):1208-12. No abstract available. PMID 5339656
- [Background] Miles DS, Gotshall RW, Golden JC, Tuuri DT, Beekman RH 3rd, Dillon T. Accuracy of electrical impedance cardiography for measuring cardiac output in children with congenital heart defects. Am J Cardiol. 1988 Mar 1;61(8):612-6. doi: 10.1016/0002-9149(88)90775-8. PMID 3344687
- [Background] Taylor K, La Rotta G, McCrindle BW, Manlhiot C, Redington A, Holtby H. A comparison of cardiac output by thoracic impedance and direct fick in children with congenital heart disease undergoing diagnostic cardiac catheterization. J Cardiothorac Vasc Anesth. 2011 Oct;25(5):776-9. doi: 10.1053/j.jvca.2011.05.002. PMID 21684761
- [Background] Fontana P, Boutellier U, Toigo M. Reliability of measurements with Innocor during exercise. Int J Sports Med. 2009 Oct;30(10):747-53. doi: 10.1055/s-0029-1225340. Epub 2009 Jul 29. PMID 19642059
- [Background] Dong L, Wang JA, Jiang CY. Validation of the use of foreign gas rebreathing method for non-invasive determination of cardiac output in heart disease patients. J Zhejiang Univ Sci B. 2005 Dec;6(12):1157-62. doi: 10.1631/jzus.2005.B1157. PMID 16358372
- [Background] Warburton DE, Haykowsky MJ, Quinney HA, Humen DP, Teo KK. Reliability and validity of measures of cardiac output during incremental to maximal aerobic exercise. Part II: Novel techniques and new advances. Sports Med. 1999 Apr;27(4):241-60. doi: 10.2165/00007256-199927040-00004. PMID 10367334
- [Background] Agostoni P, Cattadori G, Apostolo A, Contini M, Palermo P, Marenzi G, Wasserman K. Noninvasive measurement of cardiac output during exercise by inert gas rebreathing technique: a new tool for heart failure evaluation. J Am Coll Cardiol. 2005 Nov 1;46(9):1779-81. doi: 10.1016/j.jacc.2005.08.005. Epub 2005 Oct 10. No abstract available. PMID 16256885
- [Background] Gabrielsen A, Videbaek R, Schou M, Damgaard M, Kastrup J, Norsk P. Non-invasive measurement of cardiac output in heart failure patients using a new foreign gas rebreathing technique. Clin Sci (Lond). 2002 Feb;102(2):247-52. PMID 11834145
- [Background] Wiegand G, Kerst G, Baden W, Hofbeck M. Noninvasive cardiac output determination for children by the inert gas-rebreathing method. Pediatr Cardiol. 2010 Nov;31(8):1214-8. doi: 10.1007/s00246-010-9806-6. Epub 2010 Oct 13. PMID 20941596
- [Background] Wiegand G, Binder W, Ulmer H, Kaulitz R, Riethmueller J, Hofbeck M. Noninvasive cardiac output measurement at rest and during exercise in pediatric patients after interventional or surgical atrial septal defect closure. Pediatr Cardiol. 2012 Oct;33(7):1109-14. doi: 10.1007/s00246-012-0239-2. Epub 2012 Feb 22. PMID 22354224
- [Background] Marma AK, Opotowsky AR, Fromm BS, Ubeda-Tikkanen A, Porras D, Rhodes J. Noninvasive cardiac output estimation by inert gas rebreathing in pediatric and congenital heart disease. Am Heart J. 2016 Apr;174:80-8. doi: 10.1016/j.ahj.2016.01.006. Epub 2016 Jan 19. PMID 26995373
- [Background] Perrault H, Richard R, Kapchinsky S, Baril J, Bourbeau J, Taivassalo T. Addressing Assumptions for the Use of Non-invasive Cardiac Output Measurement Techniques During Exercise in COPD. COPD. 2016;13(1):75-81. doi: 10.3109/15412555.2015.1043985. Epub 2015 Sep 25. PMID 26408087
- [Derived] Filaire L, Chalard A, Perrault H, Tresorier R, Lusson JR, Pereira B, Costes F, Dauphin C, Richard R. Validation of intracardiac shunt using thoracic bioimpedance and inert gas rebreathing in adults before and after percutaneous closure of atrial septal defect in a cardiology research unit: study protocol. BMJ Open. 2019 May 27;9(5):e024389. doi: 10.1136/bmjopen-2018-024389. PMID 31133575